CLINICAL TRIAL: NCT00377143
Title: PRospective Evaluation Comparing Initiation of Warfarin StrategiEs (PRECISE): Pharmacogenetic-guided Versus Usual Care
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: similar large study planned by NHLBI
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 131-2006
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2011-09

CONDITIONS: Blood Coagulation Disorders
Keywords: warfarin; pharmacogenomic; CYP2C9; VKORC1; polymorphism, single nucleotide
MeSH Terms: conditions — Blood Coagulation Disorders; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2

INTERVENTIONS:
Drug: Warfarin Dosing

SUMMARY:
Warfarin (also called Coumadin®) is an anticoagulant drug (blood thinner) given to patients to help prevent blood clots from forming or to help prevent the growth of an existing blood clot. The purpose of this study is to collect information on a possible method used to determine the best warfarin dose for people before they start warfarin. This study will focus on finding out if a person's stable dose can be better predicted by using a new approach (called "pharmacogenetic-guided dosing") compared to the current warfarin dosing method. The pharmacogenetic-guided dosing method (the new warfarin dosing method) will use a person's specific health and genetic information to calculate a patient's warfarin dose at the beginning of warfarin treatment. The hope is that through this research, we may someday be able to use an individual's genetic information to guide the selection of their specific warfarin dose at the beginning of treatment, leading to precise warfarin dosing and less need for the current trial and error process.

DETAILED DESCRIPTION:
Warfarin is the mainstay of therapy in preventing venous thromboembolism (VTE), pulmonary embolism (PE), and subsequent morbidity and mortality. Despite its proven efficacy in reducing the advent of clot formation, patient-specific warfarin dosing is difficult to predict, with the initial dose regimen often resulting in supra- and subtherapeutic anticoagulation, and subsequently increasing patients' risk of bleeding or embolism. It has been shown that interpatient warfarin dosing variability is due in part to genetic variations found in the cytochrome P450 2C9 metabolism pathway (CYP2C9), as well as proteins involved in the coagulation cascade, most importantly vitamin K epoxide reductase complex subunit 1 (VKORC1). A recent retrospective study has shown that these two genes in addition to several clinical/demographic factors account for greater than 58% of the variation in patient-specific warfarin doses. However, there have been no studies documenting prospective use of this information in selecting an initial warfarin dose. Hypothesis: Stable therapeutic management of warfarin therapy can be more precisely achieved when patients are prospectively dosed based on a pharmacogenetic-guided dosing equation compared to usual care. Aim a: To determine if pharmacogenetic-guided dosing of warfarin is superior to usual care, when defined as the accuracy of the initial versus the stable warfarin dose. This will be assessed as the mean absolute difference in initial versus stable dose. Aim b: To determine if a stable warfarin dose is more quickly achieved using the pharmacogenetic-guided dosing equation compared to usual care. This will be assessed as time to stable dose. Aim c: To determine if pharmacogenetic-guided dosing is superior to usual care in terms of overdosing and underdosing patients. This will be assessed as the fraction of the population overdosed and the fraction of population underdosed by the two methods. We propose to evaluate a pharmacogenetic-guided dosing approach compared to usual care in the initiation of warfarin management. The selected pharmacogenetic-guided equation is a validated equation that includes both genetic and clinical factors and is relatively easy to incorporate into current clinical practice. Patients newly initiating warfarin therapy in a hospital setting will be randomized to receive either pharmacogenetic-guided or usual care, with follow-up anticoagulation management services provided by the University of Florida Health System Anticoagulation Clinic. Prospectively determining patients' stable dose has important clinical implications in today's management of warfarin therapy. Being able to predetermine a patient's stable dose upon initiation of therapy has the potential to decrease the time spent in supra- and subtherapeutic anticoagulation and reduce the number of clinic visits required to achieve a stable dose. Therefore we propose this study to test if using genotype data in determining the initial warfarin dose is more effective than usual care in predicting stable dose. If we can document the value of such an approach, this will provide the level of evidence needed to translate pharmacogenetic-guided dosing of warfarin into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Newly initiating warfarin

Exclusion Criteria:

* Previous use of warfarin
* Cancer
* Hepatic Disease
* History of alcoholism
* Diarrheal illness
* Febrile Illness
* Blood dyscrasias
* Pregnancy
* Medical plan to hold warfarin administration before stable dose is achieved (ie. for surgical intervention)
* Dementia
* Active bleed
* Aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of the initial versus the stable warfarin dose, measured as mean absolute difference in initial versus stable dose

SECONDARY OUTCOMES:
Time to stable dose
The frequency of subtherapeutic and supratherapeutic international normalized ratio (INR) measurements
The fraction of population overdosed and underdosed at warfarin initiation

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Johnson, Pharm.D., Principal Investigator — University of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States